CLINICAL TRIAL: NCT00388752
Title: Acupuncture for Post Amputation Limb Pain: A Pilot Study
Brief Title: Acupuncture for the Treatment of Phantom Limb and Residual Limb Pain After Amputation
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Walter Reed Army Medical Center (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #06-20011A
Record Dates: First submitted 2006-10-16; First posted 2006-10-17 (Estimated); Last update posted 2007-06-06 (Estimated); Status verified 2006-10

CONDITIONS: Phantom Limb; Residual Limb Pain; Traumatic Amputation; Amputation
Keywords: Acupuncture; Phantom limb pain; Residual limb pain; amputation; amputee; traumatic; surgical; Traumatic amputation upper extremity; Traumatic amputation lower extremity; Surgical amputation upper extremity; Surgical amputation lower extremity
MeSH Terms: conditions — Phantom Limb; Amputation, Traumatic | interventions — Acupuncture Therapy

INTERVENTIONS:
Procedure: Acupuncture

SUMMARY:
The purpose of this study is to identify the best treatment sequence and combination of acupuncture points for the treatment of phantom limb or residual limb pain in the traumatic/surgical amputee.

DETAILED DESCRIPTION:
The purpose of this pilot study is to identify the optimum combination of acupuncture points and treatment sequence in the treatment of post amputation limb pain in terms of the change in Phantom Limb Pain (PLP) and/or Residual Limb Pain (RLP) as measured by the Visual Analogue Scale (VAS) and the McGill Short Form Pain Questionnaire (SF-MPQ). Further, any side effects associated with the acupuncture treatment regimens, time requirements, and patient compliance with the treatment regimens will be estimated.

Study participants will be randomized to one of three acupuncture treatments: Chinese Scalp Acupuncture, French Auricular Acupuncture, or a combination of both.

ELIGIBILITY:
Inclusion Criteria:

* Amputees with traumatic/surgical amputation of a limb (greater than fingers or toes) secondary to trauma or peripheral vascular disease
* Amputees who have been cleared to begin prosthetic fitting
* Phantom and/or residual limb pain reported must be >/= 3/10
* Active duty military or dependent eligible for military benefit >/=18 years old

Exclusion Criteria:

* Congenital limb absence
* Pregnancy
* Any skin changes on the ear or scalp that would preclude placement of acupuncture needles
* Patients intubated and unable to give consent
* Patients with traumatic brain injury (TBI) diagnosed as greater than mild

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2006-09

PRIMARY OUTCOMES:
Presence/absence of phantom limb pain (PLP) and/or residual limb pain (RLP) pre/post each treatment
Level (Visual Analogue Scale [VAS]) of PLP and/or RLP pre/post each treatment
Level (VAS) of PLP and/or RLP one hour post each treatment
Presence/absence and level of PLP and/or RLP two weeks after final treatment

SECONDARY OUTCOMES:
Changes in medication regimen during treatment period and after final treatment
Changes in sleep habits during treatment period and after final treatment
Any change in phantom limb sensation (PLP) after final treatment
Length of time for each treatment
Any discomfort associated with each treatment
Overall satisfaction at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Tammy J Penhollow, D.O., Principal Investigator — Walter Reed Army Medical Center: Anesthesia & Operative Service, Dept of Surgery
Locations (1):
- Walter Reed Army Medical Center, Washington D.C., District of Columbia, United States